CLINICAL TRIAL: NCT04210674
Title: Effects of Argan Spinosa Oil in the Treatment of Diaper Dermatitis in Infants and Toddlers: A Quasi-Experimental Trial
Brief Title: Effects of Argan Spinosa Oil in the Treatment of Diaper Dermatitis in Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Nihaya Al shyab, Associate Professor of Child and Adolescent Health, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: argan oil
Record Dates: First submitted 2019-12-09; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Diaper Rash
Keywords: Argan oil; Infant; Children; Diaper Dermatitis; Topical Steroid Ointment
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Intervention Model Description: All children were randomly divided into two groups to receive either topical steroid ointment or the traditional medicinal product of Argan spinosa oil
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the treatment was distributed with sequentially numbered, sealed, and randomized envelope. The pediatrician, participant, children's caregiver and outcome assessor were not informed about the treatment code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The traditional medicinal product of Argan spinosa oil (Experimental): The researcher talked to children's caregivers, explained the study process and provided general consistent tips to the all of them, including firstly washing the affected area only with warm water, disposing the area to the fresh air and keep the area dry; secondly spreading the traditional medicinal product of Argan spinosa oil on the affected area sparingly over the lesions borders forth times per day, then diaper the baby; finally not to apply any on the affected area such as wet wipes, essence contained soaps, barrier cream or other medications during the seventh day of the trial. The home follow-up visits took place and the researcher re-evaluated diaper area using the 5- point grading scale in the first, third and seventh day of trial.
  Interventions: Other: The traditional medicinal product of Argan spinosa oil
- The conventional topical steroid ointment (Active Comparator): The researcher talked to children's caregivers, explained the study process and provided general consistent tips to the all of them, including firstly washing the affected area only with warm water, disposing the area to the fresh air and keep the area dry; secondly spreading the conventional topical steroid ointment on the affected area sparingly over the lesions borders forth times per day, then diaper the baby; finally not to apply any on the affected area such as wet wipes, essence contained soaps, barrier cream or other medications during the seventh day of the trial. The home follow-up visits took place and the researcher re-evaluated diaper area using the 5- point grading scale in the first, third and seventh day of trial.
  Interventions: Other: The traditional medicinal product of Argan spinosa oil

INTERVENTIONS:
Other: The traditional medicinal product of Argan spinosa oil — All children were randomly divided into two groups to receive either the traditional medicinal product of Argan spinosa oil or The conventional topical steroid ointment.
  Other Names: The conventional topical steroid ointment

SUMMARY:
The study hypothesized that using the traditional medicinal product of Argan spinosa oil is more effective than conventional topical steroid ointment on the speed up of the healing process and alleviation the symptoms in children with diaper dermatitis after seven consecutive days of the treatment

DETAILED DESCRIPTION:
Non-probability convenience sampling technique was used. Before the sampling started, a randomization plan was developed using the Statistical Package for the Social Sciences (SPSS).

Treatment Approach Initial and Follow up Visits The pediatrician did the initial consultation and evaluation in a private room that assured child information privacy at the baseline day in order to determine the DD severity level using the 5-point grading scale, after that he/she prescribed the treatment with sequentially numbered, sealed, and randomized envelope. The pediatrician was not informed about the bottles code, and then the researcher conducted a face-to-face interview in a private room with parents of children who were included in the study. The interviews were guided by a structured checklist were developed based on literature by the researcher. The checklist collected information regarding 27 variables that are potential, or suspected, to be associated with risk factors with DD.

The researcher talked to children's caregivers, explained the study process and provided general consistent tips to the all of them, including firstly washing the affected area only with warm water, disposing the area to the fresh air and keep the area dry; secondly spreading the prescribed trial medications on the affected area sparingly over the lesions borders forth times per day, then diaper the baby; finally not to apply any on the affected area such as wet wipes, essence contained soaps, barrier cream or other medications during the seventh day of the trial. The home follow-up visits took place and the researcher re-evaluated diaper area using the 5-point grading scale in the first, third and seventh day of trial.

Treatment Intervention Organic Argan Spinosa Oil was available in different specialist stores in Northern Jordan, the samples were produced in Pakistan, according to the certificate information of the product, the content is organic Argan Spinosa Oil and it was extracted in August 2017 from the hardcore of the fruit by a traditional hand cold-press method. The composition of the oil as shown on the bottle label was: Campesterol (0.2%), Avenasterol (4.1%), Beta-tocopherol (.1%), Gama tocopherol (86.5%), Delta tocopherol (7.0%), Alpha-tocopherol (5.5%), Spinasterol (44.4%) and Tocopherol Totaux (738 mg/kg). The oil samples were carefully handled to avoid contamination and correctly stored and maintained in brown glass sealed bottles.

Topical hydrocortisone 1% ointment was purchased from different pharmacies in Northern Jordan, the samples were produced in Jordan by Hayat Pharmaceutical Industries, according to the certificate information of the product, the content is Econazole Nitrate 1% and Triamcinolone Acetonide 0.1% and it was produced in March 2017.

All medications were randomly coded by the researcher as "A" for Argan Spinosa Oil and "B" for topical hydrocortisone 1% ointment, then provided to the assessed Pediatrician (who was not aware of the bottles cod) with sequentially numbered, sealed, and randomized. Children's Caregivers were instructed to apply sparingly to the affected areas forth times per day for both groups for planed seven consecutive days. The volume of medications was varied depending on child weight and age.

ELIGIBILITY:
Inclusion Criteria:

1. Infants/toddlers aged two years or younger
2. Diagnosed with diaper dermatitis (DD) by a paediatrician at baseline day

Exclusion Criteria:

1. Physical history of co-morbidities
2. Disorders that require special treatment (kidney disorders, malignancy, oral or genital thrush, psoriasis, on high protein diets or minerals deficiencies such as zinc deficiency)
3. Use of oral antibiotics therapy or topical non-steroidal anti-inflammatory drugs
4. Participation in another study
5. Allergic history to the active ingredients of trial medications.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Mean Changes from Baseline in diaper dermatitis severity scores using the traditional medicinal product of Argan spinosa oil versus the conventional topical steroid ointment from enrollment day, third day and at the end of seventh day of the treatment. | through consecutive seven days for each participant
  Diaper dermatitis severity scores was measured the changes using a visual analogue scale on the enrollment day, third, and seventh day of treatment from enrollment day, third day and at the end of seventh day of the treatment.
  This grading scale is used to reflect the severity level of the dermatitis according to Davis et al. 1986. Respectively, grade-0 represents healthy normal skin; grade-1 represents slight erythema of the entire diaper area with mild irritation; grade-2 for definite erythema of the diaper area totally or in localized areas, moderate irritation; grade-3 for moderate to severe erythema, with or without oozing, in a generalized pattern and associated with papules, pustules, and extreme irritation; grade-4 in cases of severe and worse erythema involving the entire diaper area associated with oozing papules, pustules, and erosion.

SECONDARY OUTCOMES:
Potential, or suspected associated risk factors with diaper dermatitis | through data collection period, an average of six months"
  Potential, or suspected to be associated risk factors with diaper dermatitis measured using a structured checklist developed by the researcher based on the literature. Factors include: the characteristics of the infants (age, gender, and weight), and mother or caregiver (age, parity, education level, job, income, nationality and home setting (rural, semi-urban and urban), type of feedings, introduction of solid foods, general state of health of the child, recent antibiotic used before the episode, type of diaper, the number of changing diaper per a day, type of wipes, skin cleansing agents, barrier cream used, frequency of bathing, bowel frequency, history of diaper dermatitis (severity level, medication used in the previous episodes, duration of episode and frequency of diaper dermatitis per month).

CONTACTS AND LOCATIONS:
Overall Officials: Eman Alsatari, MSN, Principal Investigator — Jordan University of Science and Technology
Locations (3):
- Jordan (3):
  - Al-Ramtha governmental hospital, Irbid
  - King Abdulla university hospital, Irbid
  - Princess Rahmeh hospital, Irbid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alsatari ES, AlSheyab N, D'Sa JL, Gharaibeh H, Eid S, Al-Nusour EA, Hayajneh AA. Effects of argan spinosa oil in the treatment of diaper dermatitis in infants and toddlers: A quasi-experimental study. J Taibah Univ Med Sci. 2023 May 22;18(6):1288-1298. doi: 10.1016/j.jtumed.2023.05.008. eCollection 2023 Dec. PMID 37275956

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Results (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04210674/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04210674/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan: Result of the study (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04210674/Prot_SAP_002.pdf